CLINICAL TRIAL: NCT02684409
Title: A Phase 1, Open Label, Single-Dose Safety, Pharmacokinetic, and Tolerability Study of Zecuity® in Adolescent Subjects With a History of Acute Migraine
Brief Title: Safety, Pharmacokinetic, and Tolerability Study of Zecuity® in Adolescent Subjects With a History of Acute Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROT-CL-NP101-015.01
Record Dates: First submitted 2016-02-02; First posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Acute Migraine
MeSH Terms: interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PROT-CL-NP101-015.01 (Experimental)
  Interventions: Drug: PROT-CL-NP101-015.01

INTERVENTIONS:
Drug: PROT-CL-NP101-015.01
  Other Names: Zecuity®; Sumatriptan

SUMMARY:
This will be a Phase 1, multiple center, open label, single-dose study in otherwise healthy adolescent subjects with a history of acute migraine. Subjects will each receive one Zecuity patch application. Subjects will be admitted 2 hours prior to dosing on Day 1, and will remain in the clinical unit under supervision until the last pharmacokinetic (PK) sample is obtained. Blood will be obtained at prescribed times for PK analysis and safety assessments will be performed, including adverse event monitoring, 12-lead ECG test, patch adhesion evaluations, skin irritation evaluations, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of migraine headache, with or without aura
* Subject and subject's parent or legal guardian are able to read and write English
* Subject must have a negative drug screen.
* Female subjects are eligible for participation provided they are of non-child bearing potential or if started menses; they are on a stable regimen of acceptable contraception
* Subject has one acceptable patch application site (left or right upper arm or thigh) that is relatively hair free and has no scars, tattoos, or abrasions
* Subject must have a body mass index of between the 5th and 84th percentile for age and sex
* Subject must be nonsmokers
* Subject must have not consumed alcoholic beverages, poppy seeds, grapefruit, and/or grapefruit juice within 72 hours prior to admission to the clinic

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Subject has suspected or confirmed cardiovascular disease
* Subject has a history of epilepsy or conditions associated with a lowered seizure threshold
* Subject with Raynaud's disease
* Subject has a history of basilar or hemiplegic migraines
* Subject has a current diagnosis of a major depressive disorder
* Subject has taken non-triptan serotonergic drugs including selective serotonin reuptake inhibitors(SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs, including Wellbutrin), tricyclic antidepressants (TCAs), monoamine oxidase inhibitors (MAOIs) or preparations containing St. John's Wort within 1 month prior to screening and/or is planning to start any of these medications during the study and through the End of Study visit
* Subject with a history of a significant allergy or hypersensitivity to any component of the study patch used in this study
* Subject who has any generalized skin irritation or disease including eczema, psoriasis, melanoma, acne or contact dermatitis
* Subject is positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Female subjects who are pregnant, breast feeding, or if of childbearing potential, is not using or is unwilling to use an effective form of contraception
* Subject has known history of tolerability issues with sumatriptan
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence
* Subject has participated in a clinical study within 30 days of screening or is planning to participate in another clinical study within 30 days of last study visit
* Subject is electrically sensitive (e.g., prior iontophoresis with adverse outcome related to the current delivered by the device).

  * Additional criteria apply, please contact the investigator for more information

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety- Percentage of Participants with Adverse Events | 30 days
Patch Adherence Evaluation | 4 hours
  Adhesive Scoring Code- 0 (≥ 90% adhered (essentially no lift off of the skin)) through 4 (patch detached (patch completely off the skin))
Skin Irritation Examination | 10 days
  Skin Irritation Examination Scale- 0 (no erythema) through 4 (Intense erythema with edema and blistering/erosion)
Area under the concentration versus time curve from time 0 to the last time point with measurable concentration (Ct) (AUC0-last) | 1 day
Area under the concentration versus time curve from time 0 to infinity (AUC0-∞); calculated as AUC0-last + Ct/λz2. | 1 day
Maximum observed drug concentration (Cmax) | 1 day
Time of maximum drug concentration (Tmax) | 1 day
The terminal elimination rate constant (λz); calculated using non-linear regression Analysis | 1 day
Terminal elimination half-life (t1/2); calculated as 0.693/λz2 | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals USA